CLINICAL TRIAL: NCT04235374
Title: Testing the Efficacy of FFC-AC-EIT in Patients With Alzheimer's Disease and Related Dementias
Brief Title: Implementation of Function Focused Care in Acute Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Penn State University (Other)
Responsible Party: Principal Investigator, Barbara Resnick, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00089301; R01AG065338-01 (NIH)
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Dementia; Acute Medical Event; Hospitalization
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: randomized trial with treatment and control sites. Patients are followed for 12 months. Facilities are worked with for 12 months.
Who Masked: Participant
Masking Description: Participants as hospitals will be randomized to treatment or control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFC-AC-EIT (Experimental): The stakeholder team will meet with the research nurse facilitator to review the details of the 12 month intervention and identify unit goals. The research nurse facilitator will then work with the identified champion for 10 hours weekly during months one and two and then for four hours weekly starting in month three for a total of 12 months to implement Steps 1 to 4 of FFC-AC-EIT [(1) Environment and Policy Assessments; (2) Education; (3) Establishing Patient Goals; and (4) Mentoring and Motivating of Staff, Patients and Families]. The stakeholder team will meet with the Research Nurse Facilitator monthly to review progress. In addition to monthly visits, weekly emails containing motivational Tidbits will be sent to all stakeholder team members within the cohort. The Tidbits include such things as updates about benefits of engaging patients with ADRD in physical activity while hospitalized.
  Interventions: Behavioral: FFC-AC-EIT
- Education Only (Placebo Comparator): Education Only (EO) Control Intervention: Hospitals randomized to EO will be provided with an in-service for nursing staff on function focused care in patients with ADRD by an EO Research Nurse Facilitator using our developed PowerPoint presentations in 30-minute sessions as is currently done in usual practice.
  Interventions: Behavioral: FFC-AC-EIT

INTERVENTIONS:
Behavioral: FFC-AC-EIT — The two intervention arms will receive the same educational information. The education group will not be exposed to any other activities. The FFC-AC-EIT will focus strongly on motivation of staff and patients to get the patients engaged in functional and physical activities.
  Other Names: FFC-AC-EO

SUMMARY:
Older adults with Alzheimer's Disease and Related Dementias (ADRD) comprise approximately 25% of hospitalized older adults. These individuals are at increased risk for functional decline, delirium, falls, behavioral symptoms associated with dementia (BPSD) and longer lengths of stay. Physical activity during hospitalization (e.g., mobility,bathing, dressing) has a positive impact on older adults including prevention of functional decline, less pain, less delirium, less BPSD, fewer falls, shorter length of stay and decreased unplanned hospital readmissions. Despite known benefits, physical activity is not routinely encouraged and older hospitalized patients spend over 80% of their acute care stay in bed. Challenges to increasing physical activity among older patients with ADRD include environment and policy issues (e.g., lack of access to areas to walk); lack of knowledge among nurses on how to evaluate, prevent and manage delirium and BPSD; inappropriate use of tethers; beliefs among patients, families, and nurses that bed rests helps recovery and prevents falls; and lack of motivation/willingness of patients to get out of bed. To increase physical activity and prevent functional decline while hospitalized we developed Function Focused Care for Acute Care (FFC-AC-EIT) for patients with ADRD. Implementation of FFC-AC-EIT changes how care is provided by having nurses teach, cue, and help patients with ADRD engage in physical activity during all care interactions. FFC-AC-EIT was developed using a social ecological model, social cognitive theory and the Evidence Integration Triangle. It involves a four-step approach that includes: (1) Environment and Policy Assessments; (2) Education; (3) Establishing Patient Goals; and (4) Mentoring and Motivating of Staff, Patients and Families. The purpose of this study is to test the efficacy of FFC-AC-EIT within 12 hospitals in Maryland and Pennsylvania randomized to FFC-AC-EIT or Function Focused Care Education Only (EO) with 50 patients recruited per hospital (total sample 600 patients). Aim 1 will focus on efficacy at the patient level based primarily on physical activity, function, and participation in function focused care, and secondarily on delirium, BPSD, pain, falls, use of tethers, and length of stay; and all of these outcomes (except length of stay and tethers) along with emergency room visits, re-hospitalizations and new long term care admissions at 1, 6 and 12 months post discharge; and at the unit level the aim is to evaluate the impact of FFC-AC-EIT on policies and environments that facilitate function and physical activity at 6, 12 and 18 months post implementation. Hospitals randomized to FFC-AC-EIT will be compared with those randomized to Function Focused Care Education Only (EO). Aim 2 will evaluate the feasibility, based on treatment fidelity (delivery, receipt, enactment)136, and relative cost and cost savings of FFC-AC-EIT versus EO. Findings will address several prioritized areas of research: a focus on ADRD; improving physical function; and training of hospital staff and will demonstrate efficacy of an approach to care for patients with ADRD that can be disseminated and implemented across all acute care facilities.

DETAILED DESCRIPTION:
After hospitals are recruited they will be randomized to cohort and randomly assigned to treatment so that the hospital will receive either FFC-AC-EIT or EO. FFC-AC-EIT is implemented by a Research Nurse Facilitator working with the stakeholder team and unit champions for 10 hours weekly during months one and two and then for four hours weekly starting in month three for a total of 12 months. Timing of the intervention activities will be flexible based on the needs of the unit. The first meeting with the stakeholder team will be 1-2 hours and the remaining meetings will be approximately 30 minutes monthly to update the stakeholders on progress and any challenges associated with implementation of FFC-AC-EIT. The majority of the time on the unit by the Research Nurse Facilitator will be spent with the champions helping and assuring that they are engaging staff in function focused care activities via the four steps of FFC-AC-EIT. Once hospitals are randomized we will set up a time to meet with the identified contact to determine the stakeholder team members and champions and organize the first stakeholder team meeting. The first meeting will provide an overview of the implementation of Steps 1 to 4 [(1) Environment and Policy Assessments; (2) Education; (3) Establishing Patient Goals; and (4) Mentoring and Motivating of Staff, Patients and Families] and will address the unit challenges to implementing function focused care using a Brainstorming approach. In the first two months the Research Nurse Facilitator completes the environment and policy assessments with the champions and implements appropriate changes on the units and plans and provides staff education and makes available information for patients and families/ caregivers. The education reviews function focused care. Ongoing work between the champions and the Research Nurse Facilitator focuses on motivating staff and patients to work toward achievement of patient goals and established unit goals. The stakeholder team will continue to meet with the Research Nurse Facilitator monthly (approximately 30 minutes) over the 12-month intervention period to review progress and to help champions overcome any identified multilevel challenges. In addition to monthly visits, weekly emails containing motivational Tidbits will be sent to all stakeholder team members within the cohort. The Tidbits include such things as updates about benefits of engaging patients with ADRD in physical activity while hospitalized. To further facilitate implementation we will give each treatment site: 1) a 100 dollar gift certificate from Nasco (Nasco.com) to buy supplies for the unit to engage patients with ADRD in physical activities (e.g., age-appropriate weights; soft horseshoe toss game); 2) 1000 dollars at the end of the study for each champion to attend a conference and submit an abstract focused on optimizing function and physical activity of hospitalized older adults with ADRD. Education Only (EO) Control Intervention: Hospitals randomized to EO will be provided with an in-service for nursing staff on function focused care in patients with ADRD by an EO Research Nurse Facilitator using our developed PowerPoint presentations in 30-minute sessions as is currently done in usual practice.

ELIGIBILITY:
Inclusion Criteria:

1. are admitted into the hospital from any setting during the 12 month implementation period;
2. are 55 years of age or older;
3. are admitted onto a medical unit for any medical diagnosis; and
4. screen positive for dementia based on two well-validated scales: a score of ≤ 25 on the Montreal Cognitive Assessment (MoCA) and a score of >2 on the AD8 Dementia Screening Interview; have mild to moderate stage dementia based a score of 0.5 to 2.0 on the Clinical Dementia Rating Scale (CDR); and lastly to differentiate between dementia and mild cognitive impairment eligibility is based on evidence of functional impairment with a score of 9 or greater on the Functional Activities Questionnaire (FAQ).

Exclusion Criteria:

1. are enrolled in Hospice;
2. have been on the unit for greater than 48 hours;
3. do not have a family member/caregiver that we can contact;
4. anticipate surgery; or
5. have a major acute psychiatric disorder, or significant neurological condition associated with cognition other than dementia.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Resnick, PhD, Principal Investigator — University of Maryland
Locations (14):
- United States (14):
  - Luminus Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland Baltimore Washington Medical Center, Baltimore, Maryland
  - University of Maryland Hospital, Baltimore, Maryland
  - Midtown Hospital, Baltimore, Maryland
  - University of Maryland Baltimore Washington Medical Center, Glen Burnie, Maryland
  - University of maryland Upper Chesapeake Hospital, Perryville, Maryland
  - University of Maryland Saint Joseph Medical Center, Towson, Maryland
  - Jefferson Abbington, Abington, Pennsylvania
  - Lancaster Hospital, Lancaster, Pennsylvania
  - Jefferson Lansdale, Lansdale, Pennsylvania
  - Jefferson Lansdale (control);, Philadelphia, Pennsylvania
  - Hospital University of Pennsylvania - Cedar Avenue, Philadelphia, Pennsylvania
  - Jefferson Methodist, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Resnick B, Boltz M, Galik E, Kuzmik A, McPherson R, Drazich B, Kim N, Zhu S, Wells CL. Measurement of Physical Activity Among Hospitalized Older Adults Living With Dementia. Rehabil Nurs. 2024 Jul-Aug 01;49(4):115-124. doi: 10.1097/RNJ.0000000000000464. Epub 2024 Jun 20. PMID 38904657

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: hospitals
Groups:
- FFC-AC-EIT: The stakeholder team will meet with the research nurse facilitator to review the details of the 12 month intervention and identify unit goals. The research nurse facilitator will then work with the identified champion for 10 hours weekly during months one and two and then for four hours weekly starting in month three for a total of 12 months to implement Steps 1 to 4 of Function Focused Care for Acute Care Using the Evidence Integration Triangle (FFC-AC-EIT) [(1) Environment and Policy Assessments; (2) Education; (3) Establishing Patient Goals; and (4) Mentoring and Motivating of Staff, Patients and Families]. The stakeholder team will meet with the Research Nurse Facilitator monthly to review progress. In addition to monthly visits, weekly emails containing motivational Tidbits will be sent to all stakeholder team members within the cohort. The Tidbits include such things as updates about benefits of engaging patients with Alzheimer's Disease and Related Dementia (ADRD) in physical activity while hospitalized.
  FFC-AC-EIT: The two intervention arms will receive the same educational information. The education group will not be exposed to any other activities. The FFC-AC-EIT will focus strongly on motivation of staff and patients to get the patients engaged in functional and physical activities.
Period: Overall Study
Arm/Group | FFC-AC-EIT | Education Only
Started | 220; 6 hospitals | 235; 6 hospitals
Completed | 105; 6 hospitals | 129; 6 hospitals
Not Completed | 115; 0 hospitals | 106; 0 hospitals
Not completed — Death | 91 | 91
Not completed — Refused | 2 | 2
Not completed — Unavailable | 12 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Withdrawal by Legally Authorized Representative | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- FFC-AC-EIT: treatment with the intervention FFC-AC-EIT
- Education Only: Treatment with control for attention with education only
- Total: Total of all reporting groups
Arm/Group | FFC-AC-EIT | Education Only | Total
Number analyzed (Participants) | 220 | 235 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.6 (7.8) | 81.4 (9.0) | 82.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 150 | 285
  Male | 85 | 85 | 170
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 92 | 141
  White | 162 | 135 | 297
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Barthel index [Mean (Standard Deviation); unit: units on a scale] — A measure of 10 activities of daily living with scores ranging from 0 to 100 and higher scores indicating better physical function.
  units on a scale | 49.2 (27.3) | 54.9 (27.1) | 51.5 (27.0)
The Physical Activity Survey [Mean (Standard Deviation); unit: units on a scale] — The Physical Activity Survey is a subjective measure of time spent in physical activities over 24 hours based on input from an informant. A total of 37 activities iin the following areas are included: locomotion (e.g., walking, wheelchair mobility), personal care (e.g., bathing), structured exercise (e.g., physical and occupational therapy), recreational activity (music), and repetitive behavior (moving objects repeatedly). scores range from 0 to 37 with each activity considered as done at least once during the day. Higher scores are indicative of more physical activities done.
  units on a scale | 8.2 (5.0) | 9.6 (6.0) | 8.8 (5.5)
Neuropsychiatric inventory [Mean (Standard Deviation); unit: units on a scale] | 1.4 (2.7) | 2.4 (3.2) | 1.9 (2.5)
Delirium [Mean (Standard Deviation); unit: units on a scale] | 1.5 (1.7) | 2.1 (1.8) | 1.7 (1.7)
Pain [Mean (Standard Deviation); unit: units on a scale] | .02 (.2) | .2 (.6) | .11 (.4)

OUTCOME MEASURES:

1. Primary Outcome: The Barthel Index
Description: A measure of 10 activities of daily living with scores ranging from 0 to 100 and higher scores indicating better physical function.
Time Frame: Scores at hospital admission, hospital discharge, 1,6, and 12 months post discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FFC-AC-EIT | Education Only
Number analyzed (Participants) | 220 | 235
score on a scale
  Baseline | 49.2 (27.3) | 54.9 (27.3)
  discharge | 52.0 (28.5) | 58.7 (27.6)
  one month | 58.2 (31.7) | 58.0 (30.6)
  six month | 61.1 (32.0) | 61.4 (27.3)
  12 month | 32.0 (12.1) | 30.1 (10.8)
Statistical Analysis 1: Comparison: FFC-AC-EIT vs Education Only; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = .06

2. Primary Outcome: The Physical Activity Survey
Description: The Physical Activity Survey is a subjective measure of time spent in physical activities over 24 hours based on input from an informant. A total of 37 activities iin the following areas are included: locomotion (e.g., walking, wheelchair mobility), personal care (e.g., bathing), structured exercise (e.g., physical and occupational therapy), recreational activity (music), and repetitive behavior (moving objects repeatedly). scores range from 0 to 37 with each activity considered as done at least once during the day. Higher scores are indicative of more physical activities done.
Time Frame: Baseline (hospital admission), hospital discharge (approximately 3 days),1, 6, and 12 months post discharge
Population: participants who had data collected at these time points.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | FFC-AC-EIT | Education Only
Number analyzed (Participants) | 220 | 235
score on scale
  Baseline | 8.2 (5.0) | 9.6 (6.0)
  Discharge: number analyzed (Participants) | 206 | 229
  Discharge | 9.2 (5.7) | 10.1 (6.4)
  one month: number analyzed (Participants) | 187 | 214
  one month | 13.6 (6.7) | 11.9 (5.7)
  six month: number analyzed (Participants) | 125 | 154
  six month | 13.9 (6.6) | 12.9 (4.6)
  twelve month: number analyzed (Participants) | 99 | 129
  twelve month | 13.4 (6.2) | 11.7 (4.4)
Statistical Analysis 1: Comparison: FFC-AC-EIT vs Education Only; Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = .05

3. Primary Outcome: The Short Confusion Assessment Method
Description: An assessment for evidence of delirium based on items reflective of behaviors associated with delirium. There are four areas considered: Acute onset and fluctuating course is scored as no (0) or yes (1). Inattention and disorganized thinking are each scored as "absent" (0 points), present in mild form (1 point), or present in severe form (2 points). Altered level of consciousness, is scored as alert or normal (0 points), vigilant or lethargic (1 point), and stupor or coma (2 points). Scores range from 0-7, with a higher score indicating greater severity of delirium.
Time Frame: baseline (hospital admission) ,hospital discharge (approximately 3 days), 1,6, and 12 months post discharge
Population: participants who had data collected at these time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FFC-AC-EIT | Education Only
Number analyzed (Participants) | 220 | 235
score on a scale
  Baseline | 1.5 (1.7) | 2.1 (1.8)
  Discharge: number analyzed (Participants) | 206 | 229
  Discharge | 1.2 (1.7) | 1.7 (1.6)
  One Month: number analyzed (Participants) | 187 | 214
  One Month | 2.2 (1.9) | 2.2 (1.8)
  Six month: number analyzed (Participants) | 125 | 154
  Six month | 2.1 (1.7) | 2.5 (1.9)
  twelve month: number analyzed (Participants) | 99 | 129
  twelve month | 2.1 (1.6) | 2.7 (2.0)
Statistical Analysis 1: Comparison: FFC-AC-EIT vs Education Only; Test type: Superiority; p = .05, Mixed Models Analysis; Mean Difference (Final Values) = .05

4. Primary Outcome: the Brief Neuropsychiatric Inventory
Description: Assessment of behavioral symptoms including delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, nighttime behaviors, and appetite/eating is done. The presence of each behavior is scored as present (1) or not present (0). The behaviors are then scored and range from 0 to 12. Higher scores are indicative of more behavioral and psychological symptoms associated with dementia.
Time Frame: baseline (hospital admission) , discharge (approximately 3 days),1,6, and 12 months post discharge nb
Population: Participants who had data collected at these time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FFC-AC-EIT | Education Only
Number analyzed (Participants) | 220 | 235
units on a scale
  Baseline | 1.4 (2.7) | 2.4 (3.2)
  Discharge | 1.7 (3.1) | 2.3 (3.1)
  One month: number analyzed (Participants) | 187 | 214
  One month | 6.6 (5.8) | 6.0 (5.7)
  Six month: number analyzed (Participants) | 125 | 154
  Six month | 5.7 (5.2) | 6.8 (6.1)
  twelve month: number analyzed (Participants) | 99 | 129
  twelve month | 3.0 (2.4) | 3.5 (2.6)
Statistical Analysis 1: Comparison: FFC-AC-EIT vs Education Only; Test type: Superiority; p = .05, Mixed Models Analysis; Mean Difference (Final Values) = .05

5. Primary Outcome: Pain in Advanced Dementia Scale (PAINAD)
Description: An objective measure of 5 behaviors commonly associated with pain. Each pain behavior is scored from 0 (no evidence) to 2 (persistant behavior). Scores are then summed for a total score that ranges from 0 to 10 with higher scores indicative of more pain.
Time Frame: change from baseline (hospital admission) to hospital discharge (approximately 3 days) date to change at 1,6, and 12 months post discharge
Population: participants who had data collected at these time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FFC-AC-EIT | Education Only
Number analyzed (Participants) | 220 | 235
units on a scale
  Baseline | .02 (.2) | .2 (.6)
  Discharge: number analyzed (Participants) | 206 | 229
  Discharge | .4 (1.1) | 1.2 (1.8)
  One month: number analyzed (Participants) | 187 | 214
  One month | 1.6 (1.7) | 1.2 (2.0)
  Six month: number analyzed (Participants) | 125 | 154
  Six month | 1.5 (1.6) | 1.3 (1.8)
  twelve month: number analyzed (Participants) | 99 | 129
  twelve month | 6.4 (1.7) | 6.4 (1.8)
Statistical Analysis 1: Comparison: FFC-AC-EIT vs Education Only; Test type: Superiority; p = .05, Mixed Models Analysis; Mean Difference (Final Values) = .05

ADVERSE EVENTS:
Time Frame: Over the 12 month study period
Description: Our adverse events are common occurrences in older adults and none of these were associated with the study intervention or participation in the study.
Arm/Group | FFC-AC-EIT | Education Only
All-Cause Mortality (participants affected / at risk) | 91/220 | 91/235
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/235
Other Adverse Events (participants affected / at risk) | 136/220 | 140/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FFC-AC-EIT (N=220) | Education Only (N=235)
Events associated with study intervention (General disorders) | 0 (0) | 0 (0) — There were no adverse events associated with study activities. these were older adults with chronic illnesses and had medical problems that had nothing to do with the study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FFC-AC-EIT (N=220) | Education Only (N=235)
falls (General disorders) | 78 | 96 — fall could impact multiple areas generally hip, head, ribs, wrist or pelvis
Emergency room visits (General disorders) | 118 | 115 — This could be from anything that the patient/family wanted to go to the Emergency room for. This could have been a fall, a rash, bleeding, pneumonia, flu, covid etc.
Hospitalizations (General disorders) | 99 | 80 — This could be for any of the many common events that happen with older adults living with dementia and other comorbid conditions such as pneumonia, bleeding, increased confusion, drug side effects, COVID, Flu, urinary tract infections etc.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT04235374/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT04235374/ICF_001.pdf